CLINICAL TRIAL: NCT05161507
Title: Targeted Axillary Dissection, Sentinel Biopsy, and Tumor Lesion Localization in Breast Cancer Patients Using the New Magnetic "Sentimag" Detection System
Brief Title: Magseed and Magtrace Localization for Breast Cancer
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: CHIR-07-Sentimag; 05/RVO-FNOs/2020 (Other Grant/Funding Number: University hospital Ostrava)
Record Dates: First submitted 2020-09-23; First posted 2021-12-17 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Breast Carcinoma; Breast Carcinoma Metastatic in Lymph Node
Keywords: Breast cancer; Sentinel lymph node; Super paramagnetic iron oxide; Magseed; Magtrace; Sentimag
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sentinel lymph node extirpation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-palpable breast cancer lesion: Patients with the non-palpable histologically confirmed breast cancer lesion that will undergo breast-conserving surgery and sentinel lymph node detection - the tumor lesion will be labeled with Magseed.
  Interventions: Procedure: Magseed
- Palpable breast cancer lesion: Patients with the palpable histologically confirmed breast cancer lesion that will undergo breast-conserving surgery and sentinel lymph node detection - The Magtrace will be injected preoperatively into the tumor and detected by Sentimag.
  Interventions: Procedure: Magtrace
- Axillary lymph node metastasis: Patients with the histologically confirmed breast cancer lesion with Axillary lymph node metastasis with pathologic confirmation by needle biopsy - the positive axillary lymph node lesion will be labeled with Magseed before the neoadjuvant systemic therapy.
  Interventions: Procedure: Axillary lymph node metastasis - needle biopsy

INTERVENTIONS:
Procedure: Magseed — Patients with the non-palpable histologically confirmed breast cancer lesion - the tumor lesion will be labeled with Magseed and patient will undergo breast-conserving surgery and sentinel lymph node detection with Tc99.
  Groups: Non-palpable breast cancer lesion
Procedure: Magtrace — Patients with the palpable histologically confirmed breast cancer lesion - The Magtrace will be injected preoperatively into the tumor and detected by Sentimag. Patient will undergo sentinel lymph node detection with Tc99 and Sentimag localization system with breast surgery.
  Groups: Palpable breast cancer lesion
Procedure: Axillary lymph node metastasis - needle biopsy — Patients with the histologically confirmed breast cancer lesion with Axillary lymph node metastasis with pathologic confirmation by needle biopsy - the positive axillary lymph node lesion will be labeled with Magseed before the neoadjuvant systemic therapy, and later during target axillary dissection will be performed the biopsy of labeled lymph node during breast surgery.
  Groups: Axillary lymph node metastasis

SUMMARY:
The aim of this study is to compare the efficacy of the Sentimag localization system and its tracer Magtrace, superparamagnetic iron oxide nanoparticles, as a tracer in sentinel node biopsy in breast cancer with Tc99 in a single-center prospective study. The other part of the study will be the implantation of the smallest non-radioactive seed, Magseed, in the non-palpable breast cancer lesions. Another part of the study will be the implantation of Magseed in the positive axillary lymph nodes in patients diagnosed with clinically positive lymph nodes that will receive neoadjuvant systemic therapy.

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of the Sentimag localization system and its tracer Magtrace, superparamagnetic iron oxide nanoparticles, as a tracer in sentinel node biopsy in breast cancer with Tc99 in a single-center prospective study. It also aims to follow skin discoloration after Magtrace injection and describe when and how it resolves. The Magtrace will be injected preoperatively. Sentinel node biopsy will be performed and detection rates will be recorded for both methods.

The other part of the study will be the implantation of the smallest non-radioactive seed, Magseed, in the non-palpable breast cancer lesions. Intraoperative localization of the seed is achieved with the use of the Sentimag probe.

Another part of the study will be the implantation of Magseed in the positive axillary lymph nodes in patients diagnosed with clinically positive lymph nodes that will receive neoadjuvant systemic therapy. To accurately assess the response in the breast and the axilla, it is important that both the positive lymph node/s are marked before neoadjuvant systemic therapy to be able to locate them later on. Systemic therapy can negatively impact lymphatic drainage and hence reduce the accuracy of the sentinel lymph node biopsy (SLNB). However, when SLNB is paired with the removal of the previously positive target lymph node, a technique called Targeted Axillary Dissection, the operation becomes a lot more accurate, with lower morbidity of the patients.

A part of the study is also the verification of the time stability of breast tumor labeling with Magseed in the period from the onset of neoadjuvance to the subsequent operation following the oncological pretreatment of the patient.

All patients will undergo sentinel lymph node detection also by the classic detection system with Tc99.

Patients receive the Magseed marker via ultrasound-guided injection into a lymph node or to non-palpable breast cancer lesion.

After completion of the study, patients are followed up within 6-30 days post-surgery at our surgical clinic.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cT0-4 breast cancer
* Without/ With axillary lymph node metastasis with pathologic confirmation by needle biopsy
* With/ without received neoadjuvant chemotherapy prior to surgical resection

Exclusion Criteria:

* Distant metastases
* The subject is known to be pregnant
* Pacemaker of another implantable device in the chest wall
* Allergy to dextran or other iron-containing particles

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with breast carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of Magseed placement | During the surgical procedure
  Accuracy of Magseed placement will be measured regarding its position towards the lymph node in mm. Will be defined as accurate, marginal or inadequate. Descriptive statistics will be used to summarize accuracy of placement. Other statistical methods, when appropriate, may be used for analysis.
Surgeon-rated ease of detected lymph node localization and removal | During the surgical procedure
  Descriptive statistics will be used to summarize surgeon rated ease of localization.
Number of nodes retrieved within the surgical specimen containing the Magseed | During the surgical procedure
  Descriptive statistics will be used to summarize number of nodes retrieved within the surgical specimen containing the Magseed.
Surgeon-rated ease of detected labeled lesion localization and removal | During the surgical procedure
  Descriptive statistics will be used to summarize number of nodes retrieved within the surgical specimen containing the Magseed.
Transcutaneous detection rate | During the surgical procedure
  Descriptive statistics will be used to summarize transcutaneous detection rate.
Incidence of adverse events | Up to 6 weeks post-procedure
  Toxicity data will be summarized by frequency tables. For the toxicity endpoint, per-treated analysis will be used to include any patient who received the treatment regardless of the eligibility nor the duration or dose of the treatment received.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Toman, MD, Principal Investigator — University Hospital Ostrava; Otakar Kubala, MD,PhD, Study Chair — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be made available to other researchers upon request.

REFERENCES:
- [Background] Rubio IT, Diaz-Botero S, Esgueva A, Rodriguez R, Cortadellas T, Cordoba O, Espinosa-Bravo M. The superparamagnetic iron oxide is equivalent to the Tc99 radiotracer method for identifying the sentinel lymph node in breast cancer. Eur J Surg Oncol. 2015 Jan;41(1):46-51. doi: 10.1016/j.ejso.2014.11.006. Epub 2014 Nov 15. PMID 25466980
- [Background] Greenwood HI, Wong JM, Mukhtar RA, Alvarado MD, Price ER. Feasibility of Magnetic Seeds for Preoperative Localization of Axillary Lymph Nodes in Breast Cancer Treatment. AJR Am J Roentgenol. 2019 Oct;213(4):953-957. doi: 10.2214/AJR.19.21378. Epub 2019 Jun 5. PMID 31166765
- [Background] Zacharioudakis K, Down S, Bholah Z, Lee S, Khan T, Maxwell AJ, Howe M, Harvey J. Is the future magnetic? Magseed localisation for non palpable breast cancer. A multi-centre non randomised control study. Eur J Surg Oncol. 2019 Nov;45(11):2016-2021. doi: 10.1016/j.ejso.2019.06.035. Epub 2019 Jun 26. PMID 31288944